CLINICAL TRIAL: NCT01151605
Title: The Suppression of Toll Like Receptors by Insulin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University at Buffalo (Other)
Collaborators: American Diabetes Association (Other)
Responsible Party: Principal Investigator, Paresh Dandona, MD, University at Buffalo
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1934; 708CR13 (Other Grant/Funding Number: American Diabetes Association)
Record Dates: First submitted 2010-06-25; First posted 2010-06-28 (Estimated); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Insulin Resistance
MeSH Terms: conditions — Insulin Resistance | interventions — Insulin Infusion Systems

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- obese subjects (Experimental): obese (BMI >30Kg/m2) subjects infused with insulin dextrose or saline 1 week apart. Each infusion will continue for up to 14 hr
  Interventions: Drug: insulin infusion; Drug: Dextrose infusion; Drug: Saline Infusion
- Normal weight subjects (Active Comparator): Normal weight subjects infused with insulin dextrose or saline 1 week apart. Each infusion will continue for up to 14 hr
  Interventions: Drug: insulin infusion; Drug: Dextrose infusion; Drug: Saline Infusion
- obese type 2 diabetes subjects (Experimental): obese (BMI >30Kg/m2) subjects with type 2 diabetes infused with insulin dextrose or saline 1 week apart. Each infusion will continue for up to 14 hr
  Interventions: Drug: insulin infusion; Drug: Dextrose infusion; Drug: Saline Infusion

INTERVENTIONS:
Drug: insulin infusion — insulin to be infused at 3.5 units/hour along with Dextrose 12.5% at a rate to achieve blood glucose levels between 80-120mg/dl
  Other Names: Intravenous regular insulin infusion
Drug: Dextrose infusion — Dextrose 12.5% will be infused at a rate to maintain blood glucose level 80-120mg/dl
  Other Names: Intravenous dextrose solution infusion
Drug: Saline Infusion — Saline will be infused at 100ml/hr
  Other Names: normal saline infusion

SUMMARY:
This study will help us understand the possible beneficial effects of insulin in inflammation. Inflamamtion is considered to be the cause of atherosclerosis and heart disease.

DETAILED DESCRIPTION:
Obesity and type 2 diabetes are major health problems in the United States and the world. Both conditions are characterized by increased inflammation and oxidative stress and are associated with increased risk of cardiovascular disease.

Our previous work shows that insulin exerts a prompt and powerful anti-inflammatory effect, on circulating blood cells and in plasma in healthy subjects and in critically ill patients.

Toll like receptors (TLRs) recognize bacterial and viral products like endotoxin and viruses and are major determinants of the inflammatory response against foreign pathogens. In view of the recent data showing that TLRs recognize a range of molecules and proteins that are not of pathogenic source like saturated lipids and that TLRs are involved in the pathogenesis of atherosclerosis which leads to cardiovascular disease and insulin resistance which leads to type 2 diabetes (DM) we hypothesized that insulin infusion suppresses TLRs expression.

Our preliminary data show that insulin infusion for 4 hours reduces the levels of many TLRs and thus might protect from inflammation induced conditions We therefore propose to investigate, in more detail, the effect of infusing different doses of insulin on TLRs mRNA and protein levels and its activity in obese and DM subjects over a longer infusion period and a larger number of subjects in circulating white blood cells and in fat tissue. Also we will be comparing the baseline levels of TLRs and TLRs related proteins as well as their modulation by insulin between normal, obese and DM subjects.

ELIGIBILITY:
INCLUSION CRITERIA

Lean Group:

1. Age: 20 to 65 years of age inclusive
2. Sex: male or female
3. Normal fasting plasma glucose (65-100 mg/dl)
4. Normal BMI (20-25)

Obese Group:

1. Age: 20 to 65 years of age inclusive
2. Sex: male or female
3. Normal fasting plasma glucose (65-100 mg/dl)
4. BMI> 30

DM Group:

1. Type 2 Diabetes Mellitus
2. Age: 20 to 65 years of age inclusive
3. Sex: male or female
4. BMI >30
5. Hba1c < 8%
6. If on statins, angiotensin converting enzyme inhibitor, angiotensin receptor blocker or low dose aspirin, should be on a stable dose for one month.

EXCLUSION CRITERIA

1. Pregnancy
2. Congestive heart failure
3. Heart Rate <50 beats /minute
4. Sick Sinus Syndrome
5. Second or third degree heart block
6. Blood pressure <80 mm systolic or > 160/100 mmHg
7. Coronary event or procedure (myocardial infarction, unstable angina, coronary artery bypass surgery or coronary angioplasty) in the previous three months
8. Hepatic disease (transaminase > 3 times normal)
9. Renal impairment (serum creatinine > 1.5)
10. History of drug or alcohol abuse within past one year
11. Participation in any other concurrent clinical trial
12. Potassium (K+) values <3.5 meq/l to > 5.5 meq/l)
13. Any other life-threatening, non-cardiac disease
14. Use of an investigational agent or therapeutic regimen within 30 days of study
15. Type 2 diabetics on thiazolidinediones and/ or insulin
16. Subjects on steroids, NSAIDS or antioxidants
17. Patients taking exenatide or sitaglipin or loop diuretics
18. Anemia (Hemoglobin level less than 12gm/dl in females and 13gm/dl in males) 19)Allergy to lidocaine

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2008-09 (Actual); Primary Completion 2013-09 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
The Suppression of Toll Like receptors by Insulin | 24 hours
  Expression of TLR2, TLR4, TLR7 and TLR9 mRNA in mononuclear cells and adipose tissue

SECONDARY OUTCOMES:
TLR expression | 0 hours
  Basal TLR expression in obese and type 2 diabetic subjects as compared to lean subjects

CONTACTS AND LOCATIONS:
Overall Officials: Paresh Dandona, MBBS, Principal Investigator — The Research foundation of SUNY at Buffalo
Locations (1):
- Millard Fillmore Gates Hospital, Buffalo, New York, United States